CLINICAL TRIAL: NCT03164044
Title: Improved Basophil Activation Test (BAT) in the Diagnostics of IgE-mediated Drug Allergy
Brief Title: Improved Basophil Activation Test (BAT) in the Diagnostics of Drug Allergy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Republican Research and Practical Center for Epidemiology and Microbiology (Other)
Responsible Party: Principal Investigator, Andrei Y. Hancharou, Head of the Laboratory for Immunology and Cellular Biotechnology, The Republican Research and Practical Center for Epidemiology and Microbiology
Other Study IDs: RRPCEM_BAT
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Drug Allergy; Antibiotic Allergy; NSAID-Induced Anaphylactoid Reaction
Keywords: Allergy; Drug allergy; Basophil activation test; Flow cytometry
MeSH Terms: conditions — Drug Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood drained into tubes with sodium heparin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with drug allergy: Patients with drug allergy to antibiotics or NSAIDs

SUMMARY:
Current study evaluates the use of the improved Basophil Activation Test (BAT) in the diagnostics of IgE-mediated allergy to antibiotics and non-steroidal anti-inflammatory drugs (NSAIDs).

DETAILED DESCRIPTION:
Current study evaluates the use of the improved Basophil Activation Test (BAT) in the diagnostics of IgE-mediated allergy to antibiotics and non-steroidal anti-inflammatory drugs (NSAIDs). Among commonly used CD63/CD203c markers, newly proposed molecules, such as CD69, CD107a, CD164, CD13, CD11b and CD300a will be assayed. Results obtained together with the other clinical data will be used to calculate sensitivity and specificity of the method.

ELIGIBILITY:
Inclusion Criteria:

* suspected allergy to antibiotics or NSAIDs in the last 1 year.

Exclusion Criteria:

* autoimmune diseases;
* HIV;
* hepatitis B/C;
* other acute or chronic infectious diseases;
* malignant neoplasms;
* leukemia;
* other severe acute or chronic intercurrent diseases;
* pregnancy/lactation;
* refuse of patient to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the suspected allergy to antibiotics or NSAIDs
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the improved Basophil Activation Test (BAT) in the Diagnostics of Drug Allergy | 1 month
  Sensitivity of the improved Basophil Activation Test (BAT) in the diagnostics of allergy to antibiotics or NSAIDs
Specificity of the improved Basophil Activation Test (BAT) in the Diagnostics of Drug Allergy | 1 month
  Specificity of the improved Basophil Activation Test (BAT) in the diagnostics of allergy to antibiotics or NSAIDs

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, Dr, Study Director — Laboratory for Immunology and Cellular Biotechnology, The Republican Research and Practical Center for Epidemiology and Microbiology; Iryna U Ramanava, Principal Investigator — Laboratory for Immunology and Cellular Biotechnology, The Republican Research and Practical Center for Epidemiology and Microbiology
Locations (1):
- Andrei Hancharou, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No